CLINICAL TRIAL: NCT03871985
Title: Efficacy of Intermittent Subglottic Secretion Lavage Combined With Aspiration Preventing Ventilator Associated Pneumonia in Patients With Severe Neurological Disease：A Single-center Randomized Controlled Trial
Brief Title: Efficacy of Two Intermittent Subglottic Secretion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SSD-SSLACA
Record Dates: First submitted 2019-02-19; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2018-12

CONDITIONS: Ventilator Associated Pneumonia
Keywords: ventilator-associated pneumonia; subglottic secretion drainage; endotracheal tube; length of mechanical ventilation
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavage combined with aspiration (Experimental): Intermittent subglottic secretions lavage combined with aspiration
  Interventions: Procedure: Subglottic secretion lavage combined with aspiration
- Pure aspiration (Active Comparator): Intermittent subglottic secretions aspiration
  Interventions: Procedure: Subglottic secretion aspiration

INTERVENTIONS:
Procedure: Subglottic secretion lavage combined with aspiration — Ventilator-associated pneumonia preventive measures were applied to all patients according to VAP bundle. Subglottic secretion lavage combined with aspiration was performed every 4 hours: Underwent preoxygenation before cuff pressure checking, and was maintained between 30 and 35 cmH2O. After aspirating secretions from the mouth, nose, and airway, 2-5 mL distilled sterile water was instilled through the subglottic lumen, and then the negative pressure suction device is connected with the outer opening of the side cavity of endotracheal intubation for suction with a negative pressure of 100 mmHg, and each suction was kept under 15 seconds. Repeat lavage and aspiration until the irrigation fluid is clear. After washing, cuff pressure checking and was maintained between 25 and 30 cmH2O.
  Arms: Lavage combined with aspiration
Procedure: Subglottic secretion aspiration — Ventilator-associated pneumonia preventive measures were applied to all patients according to VAP bundle. Subglottic secretion aspiration was performed every 4 hours:Underwent preoxygenation before cuff pressure checking ,and was maintained between 25 and 30 cmH2O. After aspirating secretions from the mouth, nose, and airway, the negative pressure suction device is connected with the outer opening of the side cavity of endotracheal intubation for suction with a negative pressure of 100 mmHg, and each suction was kept under 15 seconds. Repeat suction until the secretion is completely absorbed.
  Arms: Pure aspiration

SUMMARY:
The purpose of this study is to determine the efficacy of intermittent subglottic secretion lavage combined with aspiration preventing ventilator associated pneumonia in patients with severe neurological disease

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is a common and serious complication of mechanical ventilation. Many studies have shown that the accumulation of subglottic secretions above the endotracheal cuff plays an important role in the pathogenesis of VAP. Subglottic secretion drainage (SSD) has been shown to be associated with a lower incidence of VAP in previous meta-analyses. Most studies in past reported that in the group of patients in whom endotracheal tube (ETT) was used and subglottic secretion drainage was applied compared to the group without subglottic secretion drainage.Very few studies compared two different methods of SSD,such as subglottic secretion lavage combined with aspiration or pure aspiration.The tubes need frequent cleaning as they often get blocked, especially the draining duct. This may be the reason why they are not commonly applied. However,subglottic secretion lavage combined with aspiration can reduce the incidence of tube blockage.So The purpose of this study is to determine the efficacy of intermittent subglottic secretion lavage combined with aspiration preventing ventilator associated pneumonia in patients with severe neurological disease.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18 and 80 years requiring mechanical ventilation for more than 72 hours with placement of an ETT( equipped with a dorsal suction catheter for subglottic secretion drainage)

Exclusion Criteria:

* Exclusion criteria were patients endotracheal intubation was performed before admission, history of HIV, immunosuppression, leukopenia, patient refusal,and

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2019-03-15 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of ventilator-associated pneumonia | through study completion, an average of 10 months
  is pneumonia that occurs when an artificial airway is established and mechanically ventilated

SECONDARY OUTCOMES:
Incidence of draining duct blockage | through study completion, an average of 10 months
  If mucus flow stopped during subglottic suctioning with a sudden increase of the negative pressure in the proximal port of the suction suggesting a probable occlusion

OTHER OUTCOMES:
length of mechanical ventilation | through study completion, an average of 10 months
  length of mechanical ventilation
The coincidence rate between pathogens of subglottic secretions and the lower respiratory tract | through study completion, an average of 10 months
  The coincidence rate between pathogens of subglottic secretions and the lower respiratory tract